CLINICAL TRIAL: NCT04590209
Title: Clinical and Mechanistic Study of Patients With a Recent Acrosyndrome
Brief Title: Clinical and Mechanistic Study of Patients (With COVID-19 or Not) With a Recent Acrosyndrome
Acronym: ACROCOVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP200884; N° IDRCB 2020-A0181336 (Other: ANSM)
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Adult Patients With Lesions on Fingers or Toes
Keywords: SARS-CoV-2; COVID-19; Acrosyndrome; Skin lesions
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acrosyndrome (Experimental): The blood sample, skin biopsy and other biological samples will be taken from patients
  The precise description of the semiology of skin lesions, their topography, as well as the analysis of the entire skin integument and mucous, cardiac and pulmonary auscultation and neurological examination will be done as required.
  Interventions: Other: Blood sampling; Other: Skin biopsy

INTERVENTIONS:
Other: Blood sampling — Recruited patients will be subjected to 2 blood samples of 7 mL at day 0 for serological analysis and cell collection and to an additional blood sample of 7 mL at day 15 for serological analysis
Other: Skin biopsy — Recruited patients will be subjected to a single skin biopsy at day 0 for histological and transcriptomic analysis

SUMMARY:
The recent and unexpected occurrence of patients with the development of skin lesions on the hands and/ or feet has been described recently. As these cases occurred contemporaneously with the Coronavirus Disease 2019 (COVID-19) and as it was the most often occurrence of de novo frostbites, the question raised of whether there is a direct link between the occurrence of these lesions and infection of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) the responsible for CoVID-19. Indeed, mechanisms of these lesions and the precise correlation with Sars-CoV-2 remains poorly understood. Therefore, this study aim to:

1. Determine the possible link with this virus,
2. Understand the mechanisms involved in the pathogenesis of these lesions.

DETAILED DESCRIPTION:
In this study, the investigator designed a prospective interventional study in order to collect blood samples and skin lesion biopsy at significant time points in patients who present a skin lesion. The intervention in this study is limited to some blood samples and skin biopsies.

Two 7 mL tubes of blood will be collected at consultant time for essentially serological test for the SARS-CoV-2 and for analysing certain populations of white blood cells. The second additional blood sample of 7 mL will be collected around day 15 after inclusion in a dry tube to perform a serological test for SARS-CoV-2 at a distance from the onset of skin signs.

A biopsy for histological study is usually done in patients with acrosyndrome. This is why this type of biopsy will be done as a routine care of these patients. An immunohistochemical study could complete the histological explorations using an anti-coronavirus antibody if arguments in favour of SARS-CoV-2 are demonstrated. In this study, patients who accept and sign informed consent will be proposed a skin biopsy on a characteristic lesion for freezing. This biopsy can be used for transcriptomic analysis. This may allow a better understanding of the mechanisms of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Consultant for the recent occurrence of lesions on the fingers and or toes
* Having signed an informed consent
* Affiliated or entitled to a social security regime

Exclusion Criteria:

* Patients under guardianship or under curate
* Patients under state medical assistance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Detection of SARS-CoV-2 by real-time PCR and serological test | assessing change between day 0 and day 15
  SARS-CoV-2 will be tested by Polymorphism Chain Reaction (PCR) (on the first day of consultation) and serological analysis ( at day 0 and day 15 after the first consultation)

SECONDARY OUTCOMES:
Detection of SARS-CoV-2 by metagenomics analysis | Up to 2.5 months after inclusion
  Metagenomics analysis will be performed on nasopharyngeal, tonsil and perianal samples
Detection of acrosyndrome by transcriptomic analysis of skin samples | Up to 2.5 months after inclusion
  Transcriptomic analysis will be conducted with RNA extracted from frozen skin samples

CONTACTS AND LOCATIONS:
Overall Officials: Sélim Aractingi, MD, PhD, Principal Investigator — Tarnier Hospital, AP-HP; Nicolas Dupin, MD, PhD, Study Director — Tarnier Hospital, AP-HP
Locations (1):
- Department of Dermatology, Tarnier hospital, AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No